CLINICAL TRIAL: NCT02536118
Title: Micra Transcatheter Pacing System Post-Approval Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Micra Registry
Record Dates: First submitted 2015-08-17; First posted 2015-08-31 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients implanted with Micra System: Patients implanted with a Micra Transcatheter Pacing System are eligible for enrollment into the Micra PA Registry.
  Interventions: Device: Micra Transcatheter Pacing System

INTERVENTIONS:
Device: Micra Transcatheter Pacing System — The Micra system is a miniaturized single chamber pacemaker system that is delivered via catheter through the femoral vein and is implanted directly inside the right ventricle of the heart. The Micra implantable device is a self-contained, hermetically enclosed, miniaturized single chamber pacemaker. The device is fixated via four electrically inactive nitinol tines, located on the distal end of the device.
  Other Names: Micra; Micra TPS

SUMMARY:
Medtronic is sponsoring the Micra Registry to further confirm safety and effectiveness of the Micra Transcatheter Pacing System (Micra system) when used as intended, in "real-world" clinical practice, following commercial release.

The Micra Registry is conducted within Medtronic's Product Surveillance Registry.

DETAILED DESCRIPTION:
The Micra Registry is a global, prospective, observational, multi-site registry. Patients enrolled in the Micra Registry will be prospectively followed for a minimum of 9 years post-implant or until registry closure, patient death, patient exit from the registry (i.e., withdrawal of consent), or unless patient is participating in an acute performance sub-study of the Micra Registry*.

Enrolled patients will have scheduled follow-up visits at least annually or as prompted by reportable adverse events; however, all Micra system follow-up patient visits are to be reported. Therefore, if more frequent scheduled visits occur per a provider's standard care practice, those visits are reported. The total estimated registry duration is 11 years.

*Patients contributing to an acute performance sub-study of the Micra Registry do not contribute to the FDA-regulated Post-Approval Study which includes a long-term (minimum 9-year) patient follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient is intended to receive or be treated with a Micra Transcatheter Pacing System and must be enrolled prior to the TPS implant procedure

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to be implanted with a Micra system are eligible for enrollment and all patients must be consented prior to the implant. Only geographies with regulatory approval for the Micra system are eligible to enroll patients (see locations section).
  All patients enrolled and successfully implanted with a Micra system will be followed for a minimum of 9 years, unless a patient is exited from the registry due to an unavoidable reason. If a Micra system is not successfully implanted, patients will be exited from the registry unless a Micra System and/or implant procedure related event is identified, for which the patient will be followed until the event is resolved or no further actions need to be taken.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Acute complication rate | 30-days
  To estimate acute complication rate related to the Micra system and/or implant procedure.
Long-term complication free survival | 9 years
  To estimate the chronic complication free survival rate of the Micra system.

SECONDARY OUTCOMES:
Pacing impedance (ohms) and pacing threshold (volts) | Up to 9 years
  Summary statistics of electrical performance 5-years post-implant measurements will be reported.
Complications stratified by implant type | Up to 9 years
  A listing of Micra system and/or implant procedure related complications stratified by implant types including de novo implants, previous cardiac device, or co-existing hardware. The listing will include complications will be listed including device implant date, complication category, complication date, device-relatedness and seriousness.
Estimate Micra System revision rate | Up to 9 years
  Summary statistics post-implant Micra System revisions, including system explant, replacement (with and without system explant), reposition will be reported.
Estimate System Longevity | Up to 9 years
  Summary statistics regarding battery length will be reported.
Confirm the rate response operation of the Micra system | Approximately 2 years
  Analysis of treadmill testing data from patients implanted with Micra for at least 3 months. Rate response data collected in the registry will be combined with data from the FDA Investigational Device Exemption study (NCT 02004873).

OTHER OUTCOMES:
Micra System complications, pacing impedance (ohms) and pacing threshold (volts), following exposure to MR environment | Up to 9 years
  Micra System performance will be described following use in an MR environment. A listing of MRI related events, pacing impedance (ohms) and pacing threshold (volts) over time following MR exposure may be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Micra Registry Manager, Study Director — Medtronic
Locations (156):
- United States (52):
  - Birmingham, Alabama
  - Los Angeles, California
  - Redwood City, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - Safety Harbor, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Morristown, New Jersey
  - Ridgewood, New Jersey
  - Huntington, New York
  - New York, New York
  - Poughkeepsie, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - Milwaukee, Wisconsin
- Belgium (3):
  - Brussels
  - Edegem
  - Leuven
- Canada (2):
  - Kingston, Ontario
  - Montreal
- Prague, Czechia
- Denmark (4):
  - Aarhus
  - Copenhagen
  - Hillerød
  - Odense
- France (20):
  - Annecy
  - Bayonne
  - Bordeaux
  - Brest
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Grenoble
  - Lille
  - Marseille
  - Montpellier
  - Nancy
  - Nantes
  - Neuilly-sur-Seine
  - Rennes
  - Rouen
  - Saint-Denis
  - Saint-Etienne
  - Strasbourg
  - Toulouse
  - Villeurbanne
- Germany (14):
  - Aachen
  - Berlin
  - Cologne
  - Dresden
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Hanover
  - Heidelberg
  - Jena
  - Mainz
  - Münster
  - Tübingen
  - Ulm
- Greece (2):
  - Athens
  - Marousi
- Budapest, Hungary
- Reykjavik, Iceland
- Israel (3):
  - Ashkelon
  - Jerusalem
  - Ramat Gan
- Italy (7):
  - Bari
  - Bologna
  - Brescia
  - Cotignola
  - Milan
  - Pisa
  - Roma
- Japan (4):
  - Mitaka-shi, Tokyo
  - Shinagawa, Tokyo
  - Suita
  - Yokohama
- Safat, Kuwait
- Netherlands (10):
  - Amsterdam
  - Breda
  - Eindhoven
  - Enschede
  - Groningen
  - Leiden
  - Maastricht
  - Nieuwegein
  - Rotterdam
  - The Hague
- Christchurch, New Zealand
- Norway (2):
  - Bergen
  - Trondheim
- Poland (2):
  - Poznan
  - Zabrze
- Lisbon, Portugal
- Saudi Arabia (2):
  - Jeddah
  - Riyadh
- Spain (5):
  - A Coruña
  - Barcelona
  - Santiago de Compostela
  - Toledo
  - Vitoria-Gasteiz
- Uppsala, Sweden
- Switzerland (7):
  - Basel
  - Bern
  - Fribourg
  - Geneva
  - Lausanne
  - Lugano
  - Zurich
- United Kingdom (10):
  - Birmingham
  - Bristol
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Middlesbrough
  - Nottingham
  - Southampton

REFERENCES:
- [Derived] Piccini JP, Cunnane R, Steffel J, El-Chami MF, Reynolds D, Roberts PR, Soejima K, Steinwender C, Garweg C, Chinitz L, Ellis CR, Stromberg K, Fagan DH, Mont L. Development and validation of a risk score for predicting pericardial effusion in patients undergoing leadless pacemaker implantation: experience with the Micra transcatheter pacemaker. Europace. 2022 Jul 21;24(7):1119-1126. doi: 10.1093/europace/euab315. PMID 35025987
- [Derived] El-Chami MF, Garweg C, Iacopino S, Al-Samadi F, Martinez-Sande JL, Tondo C, Johansen JB, Prat XV, Piccini JP, Cha YM, Grubman E, Bordachar P, Roberts PR, Soejima K, Stromberg K, Fagan DH, Clementy N. Leadless pacemaker implant, anticoagulation status, and outcomes: Results from the Micra Transcatheter Pacing System Post-Approval Registry. Heart Rhythm. 2022 Feb;19(2):228-234. doi: 10.1016/j.hrthm.2021.10.023. Epub 2021 Oct 29. PMID 34757189
- [Derived] El-Chami MF, Shinn T, Bansal S, Martinez-Sande JL, Clementy N, Augostini R, Ravindran B, Sagi V, Ramanna H, Garweg C, Roberts PR, Soejima K, Stromberg K, Fagan DH, Zuniga N, Piccini JP. Leadless pacemaker implant with concomitant atrioventricular node ablation: Experience with the Micra transcatheter pacemaker. J Cardiovasc Electrophysiol. 2021 Mar;32(3):832-841. doi: 10.1111/jce.14881. Epub 2021 Jan 23. PMID 33428248
- [Derived] Garg A, Koneru JN, Fagan DH, Stromberg K, Padala SK, El-Chami MF, Roberts PR, Piccini JP, Cheng A, Ellenbogen KA. Morbidity and mortality in patients precluded for transvenous pacemaker implantation: Experience with a leadless pacemaker. Heart Rhythm. 2020 Dec;17(12):2056-2063. doi: 10.1016/j.hrthm.2020.07.035. Epub 2020 Aug 4. PMID 32763431
- [Derived] El-Chami MF, Al-Samadi F, Clementy N, Garweg C, Martinez-Sande JL, Piccini JP, Iacopino S, Lloyd M, Vinolas Prat X, Jacobsen MD, Ritter P, Johansen JB, Tondo C, Liu F, Fagan DH, Eakley AK, Roberts PR. Updated performance of the Micra transcatheter pacemaker in the real-world setting: A comparison to the investigational study and a transvenous historical control. Heart Rhythm. 2018 Dec;15(12):1800-1807. doi: 10.1016/j.hrthm.2018.08.005. Epub 2018 Aug 10. PMID 30103071